CLINICAL TRIAL: NCT00523601
Title: A 8-Week, Multicenter, Open-Label, Observational Study of the Efficacy of Quetiapine Fumarate (SEROQUEL) Immediate-Release Tablets in Adult Patients With Bipolar Depression
Brief Title: Quetiapine Efficacy in Bipolar Depression Study
Acronym: QUEEN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-NKR-SER-2007/2
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-04

CONDITIONS: Bipolar Depression
Keywords: Bipolar depression; quetiapine; observational; Naturalistic
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To reassure the clinical study data on Seroquel antidepressant efficacy in patients who are diagnosed as bipolar depression

ELIGIBILITY:
Inclusion Criteria:

* The patient and the patient's legal representative (if any) must understand the nature of the study and must have given written consent
* Meet DSM-IV-TR criteria for bipolar depression at the time of baseline

Exclusion Criteria:

* Since this programme intends to describe quetiapine use in routine clinical practice when prescribed as treatment of bipolar depression, there are no programme specific exclusion criteria, other than:

Or, any of the following is regarded as a criterion for exclusion from the programme:

1. Serious or unstable, medical illness. Subjects with chronic illness may be included but must be stable and otherwise physically healthy on the basis of a physical examination, medical history
2. Known intolerance for or lack of response to quetiapine, as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Woo Bahn, Study Director — AstraZeneca Korea
Locations (3):
- South Korea (3):
  - Research Site, Kyungki-do, Goyang-si
  - Research Site, Daejun, Kwangyuk-si
  - Research Site, Kyungki-do, Suwon-si